CLINICAL TRIAL: NCT00224211
Title: Effects of Homophonic Sounds on Preterm Infants
Brief Title: Music's Effects on Premature Babies.
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Michelle Meza, Dept. of Newborn Medicine
Other Study IDs: 0506007948
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2005-09

CONDITIONS: Stress; Sleep
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- I: Stable premature infants
  Interventions: Behavioral: Music

INTERVENTIONS:
Behavioral: Music

SUMMARY:
This project is being done in order to determine if the music of Mozart will have a soothing effect on premature infants while in the neonatal intensive care unit (NICU). The primary effect to be anticipated will be a reduction in heart rate from baseline, decreased motor activity from baseline, as well as an increase of time in which the babies are in quiet sleep states while the music is being played.

Upon admission, all infants in the NICU are placed on monitors that continuously track their heart rate, respiratory rate, and oxygen saturation. During our study, data will be collected from the monitors already in use. Total time of observation will be approximately 3 hours. In addition, a monitoring device called an Actiwatch will also be used. This device looks similar to a traditional wristwatch and will be loosely strapped to the ankle or wrist of each infant using a foam and velcro strap. This device continuously monitors the baby's movements allowing us to determine if there is a change in the baby's activity level while the music is being played. It will record the baby's activity prior to the start of the music and will continue until 30 minutes after the music has stopped.

The music of Mozart will be played using a small speaker in the baby's isolette. The volume of the music will be set at 10 decibels over background noise, which on previous measurement has been found to be approximately 55 decibels (about the same as a running refrigerator or as the sound of rainfall; 60 decibels is the volume of normal conversation). The volume in the crib will be continuously monitored throughout the hour. As a final recording device, we will also intermittently be using video to capture the reactions of these infants to the music. The study will be done once a week per infant on the same day and at the same time every week

ELIGIBILITY:
Inclusion Criteria:

* All infants born at 28 weeks gestation or who are at least 28 weeks corrected age are eligible to participate. Only those in isolettes (incubators) will be included. Once a baby has been transitioned to a bassinet or crib, the baby will be pulled from the study. In order to be included, these infants must be in stable condition (without serious active medical issues) as decided by their doctor and must be breathing without the use of a ventilator.

Exclusion Criteria:

* Exclusion criteria will include a history of intraventricular hemorrhage involving the white matter (as diagnosed by head ultrasound), as well as those infants born with severe congenital deformities.

Ages: 1 Week to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Premature infants
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Meza, MD, Principal Investigator — New York Presbyterian Hospital Weill Cornell
Locations (1):
- New York Presbyterian Hospital Weill Cornell, New York, New York, United States

REFERENCES:
- [Background] Dobson R. Doctors will test whether Mozart can reduce stress in babies. BMJ. 2006 Mar 25;332(7543):688. doi: 10.1136/bmj.332.7543.688-a. No abstract available. PMID 16565122